CLINICAL TRIAL: NCT05049525
Title: Evaluation of the Response of Itraconazole and Terbinafine Therapy in Subjects With Crohn's Disease Not Responding Adequately to Current Therapy
Brief Title: Evaluation of the Response of Itraconazole and Terbinafine Therapy in Subjects With Crohn's Disease
Acronym: CD-IT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient patient enrollment
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHICC-2019-001
Record Dates: First submitted 2021-08-25; First posted 2021-09-20 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Crohn's Disease; Inflammatory Bowel Diseases
Keywords: Endoscopy; Radiology; Itraconazole; Terbinafine; Chronic Inflammatory Disorder; Malassezia Restricta
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Itraconazole; Terbinafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Itraconazole and Terbinafine (Active Comparator): During the first 4 weeks itraconazole will be administered alone at 200 mg twice daily, followed by itraconazole 200 mg twice daily and terbinafine 250 mg twice daily for the remaining 16 weeks. Both drugs will be administered orally.
  Interventions: Drug: Itraconazole 400 mg/day and terbinafine 500 mg/day administered orally.
- Placebo (Placebo Comparator): During the first 4 weeks a placebo will be administered alone at 200 mg twice daily, followed by placebo 200 mg twice daily and another placebo 250 mg twice daily for the remaining 16 weeks. Both placebos will be administered orally.
  Interventions: Drug: Itraconazole's matching placebo 400 mg/day and terbinafine's matching placebo 500 mg/day administered orally.

INTERVENTIONS:
Drug: Itraconazole 400 mg/day and terbinafine 500 mg/day administered orally. — Itraconazole capsules of 100 mg, antifungal agent. Terbinafine tablets 250 mg (as terbinafine hydrochloride), antifungal agent.
  Arms: Itraconazole and Terbinafine
Drug: Itraconazole's matching placebo 400 mg/day and terbinafine's matching placebo 500 mg/day administered orally. — Matching placebo of itraconazole capsules of 100 mg, antifungal agent. Matching placebo of terbinafine tablets 250 mg, antifungal agent.
  Arms: Placebo

SUMMARY:
This study will evaluate the response of itraconazole and terbinafine therapy compared to placebo in patients with mild to moderate Crohn's disease (CD).

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebocontrolled, phase II, proof of concept study will randomize 68 subjects at 2 to 5 clinical sites in Canada. Following signature of informed consent, subjects who meet entry criteria will be randomized in a 1:1 ratio to receive either itraconazole and terbinafine, or matching placebos. During the first 4 weeks subjects will receive itraconazole 200 mg twice daily or matching placebo, followed by itraconazole 200 mg twice daily and terbinafine 250 mg twice daily or matching placebos for the remaining 16 weeks. The 2 drugs will be administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with endoscopy/radiology confirmation of active disease within 6 months prior to enrolment;
* Mild to moderate active CD defined by the HBI score of ≥ 5 to ≤ 16 at baseline;
* Female of childbearing potential must have a negative urine pregnancy test at screening and at randomization baseline Visit 2. Women are considered not of childbearing potential if they either:
* Have had a hysterectomy or tubal ligation prior to baseline visit or;
* Are postmenopausal defined as no menses for 12 months or a FSH level (if available) in the menopausal range.
* Women of childbearing potential must agree to use an effective double method of birth control throughout the study: barrier method (e.g. male or female condoms, spermicides, sponges, foams, jellies, and diaphragm) in combination with other methods of contraception including implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, abstinence, or a sterile sexual partner.
* Subjects with the capacity to provide informed consent.

Exclusion Criteria:

* Subject with a current diagnosis of ulcerative colitis (UC);
* Contraindication to the use of itraconazole including congestive heart failure, ventricular dysfunction, ventricular arrhythmia, or negative inotropic state;
* Subjects with elevated or abnormal liver enzymes (ALT/AST>3 ULN) or patients with pre-existing chronic or active liver disease at screening;
* Female subject who is pregnant, planning to become pregnant during the study, or breastfeeding;
* Subject with renal impairment (creatinine clearance ≤ 50 mL/min using Cockcroft-Gault equation);
* Subject with a known hypersensitivity to itraconazole, terbinafine, or any of their excipients;
* Subjects on medications which interact with itraconazole: methadone, pimozide, quinidine or other CYP3A4 inhibitors;
* Positive C. difficile toxin test at screening;
* Use of steroid greater than 20 mg/day;
* Change of steroid dosage in the 2 weeks prior to enrolment;
* Change in CD therapy:

  * The Anti-TNFs, anti-integrins, anti-IL12/23 in the 4 months prior to enrolment;
  * Thiopurines or methotrexate (MTX), in the 2 months prior to enrolment;
* Participation in other clinical trial within 30 days of signing the Information and Consent Form (ICF).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the response of itraconazole and terbinafine therapy compared to placebo in subjects with CD, assessed by the Modified Harvey Bradshaw Index (HBI). | 20 Weeks
  Clinical response defined as a decrease from baseline to end of treatment in HBI ≥ 3 points

SECONDARY OUTCOMES:
To evaluate the response of the itraconazole and terbinafine therapy compared to placebo in subjects with CD on clinical remission assessed by the HBI. | 20 Weeks
  * Persistence of clinical response defined as a decrease from baseline to 8 weeks post end of treatment in HBI ≥ 3 points
  * Clinical remission defined as an HBI at end of treatment ≤ 4 points
  * Persistence of clinical remission defined as an HBI at 8 weeks post end of treatment ≤ 4 points
  * Change from baseline to end of treatment in HBI
To evaluate the response of the itraconazole and terbinafine therapy compared to placebo in subjects with CD on endoscopic response assessed by the Simplified Endoscopic Score for Crohn's disease (SES-CD). | 20 Weeks
  * Endoscopic response defined a decrease from baseline to end of treatment in SES-CD ≥ 50% of the baseline SES-CD
  * Change from baseline to end of treatment in SES-CD
To evaluate the response of the itraconazole and terbinafine therapy compared to placebo in subjects with CD on fecal and serologic markers. | 20 Weeks
  * Change from baseline to end of treatment in FC levels
  * Change from baseline to end of treatment in CRP levels
To evaluate the effect of study treatment on the primary endpoint in the subgroup of patients with positive ASCA (as measured on frozen plasma samples at end of the study). | 20 weeks
  * Change from baseline to end of treatment in ASCA levels
  * Change from baseline to 8 weeks post end of treatment in ASCA levels

OTHER OUTCOMES:
Exploratory analyses using genetic data (pharmacogenomic and metagenomics) as well as microbiotic testing will be described at a later time point and in a separate document. | 28 Weeks
  To determine the link between genetics and the response to therapy and inflammation. The microbiote genes will also be evaluated.
To evaluate steroid use between active and placebo groups at study completion. | 28 Weeks
  Steroid Use in Subjects with Crohn's Disease will be reported as the proportion of subjects who's steroid use was decreased. increased, changed or stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute (MHI); Edmond-Jean Bernard, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (4):
- Canada (4):
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No